CLINICAL TRIAL: NCT04432818
Title: Digital Life Coaching in Multiple Myeloma Patients Undergoing Hematopoietic Stem Cell Transplantation
Brief Title: Digital Life Coaching for Myeloma Patients Undergoing Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20252; NCI-2020-04166 (Other: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Digital life coaching; Hematopoietic stem cell transplantation
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pack Health's digital life coaching (DLC) (Experimental): Access to the DLC platform during a 16-week period encompassing pre-HCT conditioning chemotherapy, post-HCT recovery, and 100-day follow-up
  Interventions: Behavioral: Pack Health's digital life coaching (DLC)

INTERVENTIONS:
Behavioral: Pack Health's digital life coaching (DLC) — Pack Health smartphone-based DLC platform will be provided for 16-week subscription which allows unlimited bidirectional communication between enrolled participants and their life coach

SUMMARY:
This is the first study of digital life coaching (DLC) to engage patients during the peri-HCT period that is punctuated by intensive life changes. DLC may circumvent these limitations by combining the integrative cross-dimensional nature of life coaching with the advantages of mobile health technology. The purpose of this study is to evaluate whether ongoing participant engagement with a DLC platform is feasible for multiple myeloma (MM) patients actively undergoing hematopoietic stem cell transplantation (HCT).

DETAILED DESCRIPTION:
Participants will receive unlimited access to Pack Health's DLC platform during a 16-week period encompassing pre-HCT conditioning chemotherapy, post-HCT recovery, and 100-day follow-up. Participants will engage with Pack Health's DLC platform and complete quality of life assessments for 16 weeks beginning from enrollment. At the conclusion of the treatment period, participants will be asked to rate their satisfaction with the DLC platform

Primary Objective:

To evaluate the rate of ongoing participant engagement with a DLC platform during the study period

Secondary Objectives:

* To assess quality of life among participants during the study period
* To assess psychosocial distress among participants during the study period
* To assess sleep disturbances among participants during the study period
* To assess participant satisfaction with the DLC platform at the end of the study period

Exploratory Objectives:

* To assess benzodiazepine and zolpidem-class drug usage for anxiety or insomnia among participants during the study period
* To assess communications with treatment teams among participants during the study period
* To assess 100-day clinical outcomes among participants at the end of the study period

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of one of the following (all referred to as MM in this protocol):

  * Multiple myeloma (ICD-10 code: C90.0)
  * Extramedullary plasmacytoma (ICD-10 code: C90.2)
* Planned receipt of autologous HCT at our institution

  * Patients undergoing outpatient HCT will be eligible
  * Patients who received chemomobilization will be eligible
* Age ≥ 18, as life coaches employed by the DLC vendor are not currently trained to work with pediatric patients

Exclusion Criteria:

* Prior autologous HCT for any indication
* Physician-assessed lack of sufficient English proficiency
* Lack of ownership of a personal smartphone
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with participant's safety, provision of informed consent, or compliance with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Number of participants displaying ongoing engagement with DLC | Up to 16 weeks
  Ongoing participant engagement is defined as at least 4 or more participant-initiated interactions with the DLC platform, including at least 1 interaction in each of four 4-week study sub-periods

SECONDARY OUTCOMES:
Median PRO Measurement Information System (PROMIS) Global Health (GH) Score | Up to 16 weeks
  The PROMIS GH instrument v1.2 will be used to assess quality of life. This 10-item inventory with scores ranging from 1 to 5 with higher scores indicating a a greater quality of life. Raw PROMIS scores will subsequently be transformed to T-score metrics as per the scoring manual to reflect a population mean of 50 and standard deviation of 10. Among cancer patients, a T-score change of 5 points on any PROMIS inventory is generally considered to be clinically meaningful.
Median National Comprehensive Cancer Network (NCCN) Distress Thermometer (DT) Score | Up to 16 weeks
  The NCCN DT will be used to assess psychosocial distress. This single-item inventory uses a graphic of a thermometer to allow patients to assess their overall distress on a scale of 0=No Distress to 10= Extreme distress. The NCCN considers a cutoff score of 4 to differentiate clinically significant distress.
Median PROMIS Sleep Disturbance (SD) Short Form (SF) 4a Score | Up to 16 weeks
  The PROMIS SD SF 4a inventory will be used to measure overall sleep disturbance in past 7 days. This assessment consists of 4 items which measure sleep quality and sleep disturbances using a 5 point likert scale ranging in value from 1 to 5 with higher scores indicating greater sleep quality. Raw PROMIS scores will subsequently be transformed to T-score metrics as per the scoring manual to reflect a population mean of 50 and standard deviation of 10. Among cancer patients, a T-score change of 5 points on any PROMIS inventory is generally considered to be clinically meaningful
Median Participant Satisfaction Score | Up to 16 weeks
  Participants will be asked to provide a response, on a scale from 0 (not at all likely) to 10 (extremely likely), to the following single question: "How likely are you to recommend this life coaching tool to other patients undergoing stem cell transplantation?"

CONTACTS AND LOCATIONS:
Overall Officials: Rahul Banerjee, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banerjee R, Huang CY, Dunn L, Knoche J, Ryan C, Brassil K, Jackson L, Patel D, Lo M, Arora S, Wong SW, Wolf J, Martin Iii T, Dhruva A, Shah N. Digital Life Coaching During Stem Cell Transplantation: Development and Usability Study. JMIR Form Res. 2022 Mar 4;6(3):e33701. doi: 10.2196/33701. PMID 35039279